CLINICAL TRIAL: NCT03631602
Title: Posaconazole Oral Suspension and Itraconazole Oral Solution in Preventing Invasive Fungal Disease (IFD) in Patients With Hematopoietic Stem Cell Transplantation
Brief Title: Posaconazole vs Itraconazole in Preventing IFD Post-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, Prof.M.D.Ph.D, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Posa-SCT-01
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: IFD Post-HSCT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): posaconazole oral suspension
  Interventions: Drug: antifungal prophylaxis
- Arm 2 (Active Comparator): itraconazole oral solution
  Interventions: Drug: antifungal prophylaxis

INTERVENTIONS:
Drug: antifungal prophylaxis — posaconazole oral suspension vs itraconazole oral solution

SUMMARY:
Invasive Fungal Disease (IFD) after haematopoietic stem cell transplantation (HSCT) remain a clinical challenge.The studay aims to compare the efficacy and safety of posaconazole oral suspension vs itraconazole oral solution in preventing IFD post-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent Aged ≥13 years Patients undergoing hematopoietic stem cell transplantation. Cardiac: Left ventricular ejection fraction ≥ 50% Adequate renal and hepatic function Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females Any co-morbidity precluding the administration ofposaconazole or itraconazole

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of breakthrough IFD | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year
treatment-related mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China